CLINICAL TRIAL: NCT00853697
Title: Phase II Trial of Exogenous Testosterone Plus Dutasteride for the Treatment of Castrate Metastatic Prostate Cancer
Brief Title: Exogenous Testosterone Plus Dutasteride for the Treatment of Castrate Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: GlaxoSmithKline (Industry); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-008
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer; Castration-resistant, Metastatic
Keywords: Prostate; DUTASTERIDE; TESTOSTERONE; 09-008; Consortium Protocol LOI# c09-028
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Testosterone; Comprehensive Metabolic Panel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- testosterone with the 5α-reductase inhibitor dutast (Experimental): This trial is a multi-center, open-label, phase II trial of the combination of exogenous testosterone (AndroGel®) with the 5α-reductase inhibitor dutasteride in patients with castration-resistant metastatic prostate cancer.
  Interventions: Other: testosterone (AndroGel®) with the 5α-reductase inhibitor dutasteride

INTERVENTIONS:
Other: testosterone (AndroGel®) with the 5α-reductase inhibitor dutasteride — Patients will be treated with dutasteride 3.5 mg once daily (oral administration). To avoid rapid conversion of testosterone to DHT in case 5α-reductase is not adequately inhibited during the first few days of concurrent treatment with dutasteride and testosterone, daily dutasteride treatment will be initiated 7 days prior to testosterone initiation.
  Patients will receive AndroGel® at the dose of 15 g (3 times the standard replacement dose for hypogonadism) once daily (topical administration), starting on Day 8 and continuing for 12 weeks (or until disease progression or withdrawal from the study).
  Other Names: Patients will be seen in clinic on day 8 and then on day 15±3, day 22±3, day 36±3 and; during weeks 9 and 13 (±3 days), for a physical examination, safety assessments,; and laboratory studies. Blood will be drawn at baseline, on day 8 and then on; day 22±3, day 36±3 and during weeks 9 and 13 (±3 days), and at the completion; of the study (week 13 or if patient is removed from study earlier) for the; following assessments: CBC, comprehensive metabolic panel, PSA, testosterone,; free testosterone, DHT, SHBG, LDH, lipid panel.

SUMMARY:
Usually, the male hormone testosterone makes prostate cancer cells grow. Lowering testosterone usually stops the growth of prostate cancer. However, after a period of time without testosterone, prostate cancer cells learn to grow again.

You are able to join this trial because your prostate cancer is growing even though you have very low levels of testosterone. Studies have shown that high doses of testosterone, in this situation, can cause prostate cancer cells to stop growing.

The investigators did a study several years ago in which the investigators gave high doses of testosterone to patients such as yourself. The investigators showed that giving testosterone in this situation was safe. The investigators also showed that the investigators could, in some cases, make the PSA go down using high-dose testosterone.

The investigators believe that they can improve this type of treatment by combining testosterone with another drug called dutasteride. Dutasteride is another type of hormone. It should make testosterone levels rise. The investigators believe that combination of dutasteride and testosterone will be more a more powerful regimen against your cancer than testosterone alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have histologically confirmed castration-resistant metastatic prostate cancer with evidence of disease progression. Patients must have been in a castrate state either by orchiectomy or by GnRH analogues for a minimum of one year. In detail, they should meet all of the following criteria:
* Adult male > or = to 18 years of age
* Histologically confirmed prostate cancer, currently with progressive disease, defined as rising PSA (50% or more increase to a level of 2 ng/mL or more, based on at least 3 PSA determinations obtained at least 1 weeks apart), or 2 new osseous lesions by bone scan, soft tissue disease progression by RECIST 1.1 criteria , or the appearance of new sites of disease (by MRI/CT).
* Evidence of metastatic disease, documented within 4 weeks prior to dutasteride treatment initiation, based on a:

  * CT or MRI of the abdomen and pelvis, and/or
  * Radionuclide bone scan (in case of findings suspicious for spinal metastasis, MRI of the spine will be performed to rule out epidural disease)
* Serum PSA ≥ 2 ng/mL within 4 weeks prior to dutasteride treatment initiation in order to register to the protocol
* Normal organ function with acceptable initial laboratory values documented within 4 weeks prior to dutasteride treatment initiation:

  * WBC > or = to 3000/µL
  * Platelets > or = to 100,000/µL
  * Creatinine < or = to 2 mg/dL
  * Bilirubin < or = to 1.5 X ULN (institutional upper limits of normal)
  * AST/ALT < or = to 2 X ULN
* Karnofsky performance status > or = to 70%
* Willingness to undergo serial blood draws for the purpose of measuring CTCs and other biomarkers. MSKCC patients will need to agree to participate in MSKCC protocol 90-040 Molecular studies and clinical correlations in human prostate cancer [PI: Scher]. Also, MSKCC patients will undergo serial imaging by FDHT and FDG PET scans, under protocol 00-095 [18f]-fluoro-2-deoxy-D-glucose and [18f]-dihydro-testosterone PET imaging in patients with progressive prostate cancer (PI: Morris), depending on tracer and scanner time availability. If the study is opened in other centers outside MSKCC, those centers will be exempt from procedures linked to the MSKCC Protocol # 00-095.
* ADT treatment for at least 12 months prior to study entry with serum testosterone < 50 ng/dL.
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patients meeting any of the following criteria will not be eligible for study entry:
* Evidence of small-cell or neuroendocrine pathologic features
* Uncontrolled urinary obstruction
* Osseous metastatic disease with imminent risk (at the discretion of the treating physician) of pathologic fracture or cord compression (in patients with known spinal metastasis raising concern for cord compression, MRI of the spine should be performed to rule out epidural disease)
* Any situation where, at the discretion of the treating physician, a potential "tumor flare" would be life-threatening
* Sleep apnea (unless under good control with current treatment)
* Polycythemia vera
* History of allergic reactions attributed to compounds of similar chemical or biological composition to dutasteride
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness or social situation that would compromise compliance with study requirements
* Currently active secondary malignancy (as determined by the treating physician) other than non-melanoma skin cancer
* Use of the following medications will be prohibited during the study:

  * Current and/or previous use of the following medications:
  * Finasteride (Proscar, Propecia) or dutasteride (GI198745, Avodart) exposure within 6 months of study entry.
  * Anabolic androgenic steroids, including but not limited to testosterone, 17β testosterone esters, methyltestosterone, stanozolol, and danazol (within 6 months of study entry). Corticosteroids, including hydrocortisone, dexamethasone and prednisone are acceptable.
  * Additional hormonal therapy within 4 weeks of study entry:
  * Including megestrol, medroxyprogesterone, cyproterone, and DES
  * Drugs with antiandrogenic properties (eg, spironolactone if > 50mg/d, flutamide, bicalutamide, nilutamide, ketoconazole,* progestational agents) * Includes topical ketoconazole.
* Evidence of epidural disease by MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
determine anti-tumor effects of the combination of testosterone + dutasteride in pts with castration-resistant prostate ca, as indicated by the proportion of pts remaining alive & progression free | 12 weeks from the start of testosterone treatment

SECONDARY OUTCOMES:
To explore the association between AR expression in CRPC, as determined at baseline separately by AR FISH (performed on CTCs) and by 18F-FDHT uptake on PET scan, and progression free survival to the combination of testosterone plus dutasteride. | 12 weeks
To correlate post-treatment changes in CTCs and FDG and FDHT PET scans with post-treatment alterations in PSA and standard CT (or MRI) and bone scans. | post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org